CLINICAL TRIAL: NCT04603820
Title: An Ambispective Observational Registry Study of Pregnancy and Breast Cancer
Brief Title: Registry Study of Pregnancy and Breast Cancer
Acronym: EMBARCAM
Status: Active, not recruiting | Type: Observational
Sponsor: Spanish Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: GEICAM/2017-07
Record Dates: First submitted 2020-06-10; First posted 2020-10-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer and Pregnancy
Keywords: Pregnancy; Gestational breast cancer; Fertility preservation technique; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — A whole blood sample will be collected from all patients enrolled preferably at the enrollment visit (after signing the ICF).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An ambispective observational registry study of pregnancy and breast cancer

DETAILED DESCRIPTION:
A multicenter, observational, non-post-marketing (non-PMS), ambispective (retrospective and prospective from the registry opening) study which will enroll patients with breast cancer in any of these three situations:

1. Patients with gestational breast cancer, defined as breast cancer diagnosed during pregnancy, breastfeeding or up to a year after delivery.
2. Patients who become pregnant after a breast cancer diagnosis.
3. Patients with breast cancer who have followed any fertility preservation technique prior to the start of breast cancer treatment.

It is estimated a minimum recruitment period of approximately 3 years from the study activation. The study will remain open as long as possible in order to collect as much information as possible. GEICAM will actively search for funding for this.

Patients may also be concurrently enrolled in an interventional clinical trial. This observational registry study of pregnancy and breast cancer that collects significant data obtained from standard clinical practice, regarding the clinical characteristics of patients with breast cancer in any of the three situations described above. These data will allow the performance of both descriptive and exploratory analyses in order to evaluate the associations between different breast cancer subtypes and risk factors observed.

Finally, this study will collect high quality molecular data derived from the analysis of biological samples (paraffin-embedded tumor and peripheral blood samples) to reach a better understanding of the biological mechanisms involved in breast cancer in relation to pregnancy.

No treatment regimen will be protocol specified. This is an observational study in which clinical decisions concerning the optimum management strategy for a particular patient are taken independently of and/or prior to, any decision by the physician to invite a patient to participate in the study. The treating physician will make all treatment decisions according to his/her regular clinical practice independent of this study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient should have signed and dated the informed consent form (ICF). The enrollment of patients who have died is allowed.
2. Women aged ≥ 18 years.
3. Patients in one of the following situations:

   * Patients with breast cancer diagnosis during pregnancy, breastfeeding or within the year after delivery.
   * Patients with breast cancer who become pregnant after treatment.
   * Patients with breast cancer who were subjected to any fertility preservation method prior to the start of breast cancer treatment.
4. The patients referred to in the previous section and the patients who meet these characteristics prospectively could be enrolled retrospectively upon registry opening.
5. All cases diagnosed at the same site may be included. In order to prevent duplications, in case the patient followed her treatment and follow-up at another site, she will be enrolled as per the site where the diagnosis was made, requesting information of the treatment and progression, when possible.
6. Availability of clinical, epidemiological and progress data.

Exclusion Criteria:

Patients who do not wish to participate in the study for any reason could not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer in any of these three situations:
  1. Patients with gestational breast cancer, defined as breast cancer diagnosed during pregnancy, breastfeeding or up to a year after delivery.
  2. Patients who become pregnant after a breast cancer diagnosis.
  3. Patients with breast cancer who have followed any fertility preservation technique prior to the start of breast cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 866 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with breast cancer diagnosis during the gestation, breastfeeding, first year after the delivery (not during breastfeeding period), after a pregnancy and followed by any fertility preservation method before the anticancer treatment | Baseline visit
  Data for this study will be recorded into the electronic case report form (eCRF) via web using Remote Data Capture (RDC) from Oracle Clinical®. Once patient has signed the ICF or verified that the data of deceased patients can be included, designated site personnel will complete the register of each patient in the eCRF, where an identification number will automatically be assigned.
  Data will be recorded in the eCRF at the time of patient enrollment and approximately every year.
Race of participants with breast cancer diagnosis during the gestation, breastfeeding, first year after the delivery (not during breastfeeding period), after a pregnancy and followed by any fertility preservation method before the anticancer treatment | Baseline visit
  Data for this study will be recorded into the eCRF via web using RDC (Remote Data Capture) from Oracle Clinical®. Once patient has signed the ICF or verified that the data of deceased patients can be included, designated site personnel will complete the register of each patient in the eCRF, where an identification number will automatically be assigned.
  Data will be recorded in the eCRF at the time of patient enrollment and approximately every year.
Age of participants with breast cancer diagnosis during the gestation, breastfeeding, first year after the delivery (not during breastfeeding period), after a pregnancy and followed by any fertility preservation method before the anticancer treatment | Baseline visit
  Data for this study will be recorded into the eCRF via web using RDC (Remote Data Capture) from Oracle Clinical®. Once patient has signed the ICF or verified that the data of deceased patients can be included, designated site personnel will complete the register of each patient in the eCRF, where an identification number will automatically be assigned.
  Data will be recorded in the eCRF at the time of patient enrollment and approximately every year.

SECONDARY OUTCOMES:
Clinicopathological characteristics of cancer: Tumor size | 3 years
  Assess the clinicopathological characteristics of cancer in the patients enrolled in the study. For this, it is used the Tumor, Node, Metastasis (TNM) staging system is the most common way that doctors stage breast cancer. Patient scans and tests give some information about the stage of the cancer.
  Tumor (T) size describes the size of the tumour. Larger T is associated with inferior survival.
  Tumor cannot be assessed (TX): can't be assessed. Tis: ductal carcinoma in situ. T1: tumour is 2 centimetres (cm) across or less. T1mi: tumour is 0.1cm across or less T1a: tumour >0.1 cm but <0.5 cm T1b: tumour >0.5 cm but <1 cm T1c: tumour >1 cm but <2 cm T2: tumour >2 cm but <5 cm across. T3: tumour >5 cm across. T4a: tumour has spread into the chest wall T4b: tumour has spread into the skin and the breast might be swollen T4c: tumour has spread to both the skin and the chest wall T4d: inflammatory carcinoma
Clinicopathological characteristics of cancer: lymph node condition | 3 years
  Assess the clinicopathological characteristics of cancer in the patients enrolled in the study. For this, it is used the Tumor, Node, Metastasis (TNM) staging system is the most common way that doctors stage breast cancer. Patient scans and tests give some information about the stage of the cancer.
  Lymph Node (N) conditions describes whether the cancer has spread to the Lymph Nodes (LN). Prognosis is better when cancer has not spread to the LN. The more LN that contain cancer, the poorer prognosis tends to be.
  Node cannot be assessed (NX): LN can't be assessed N0: no Cancer Cells (CC) N1: CC in the LN in the armpit but the nodes are not stuck to surrounding tissues.
  N2a: CC in the LN in the armpit, which are stuck to each other and to other structures.
  N2b: CC in the LN behind the breast bone. N3a: CC in LN below the collarbone. N3b: CC in LN in the armpit and behind the breastbone. N3c: CC in LN above the collarbone.
Clinicopathological characteristics of cancer: metastasis presence | 3 years
  Assess the clinicopathological characteristics of cancer in the patients enrolled in the study. For this, it is used the Tumor, Node, Metastasis (TNM) staging system is the most common way that doctors stage breast cancer. Patient scans and tests give some information about the stage of the cancer.
  Metastasis (M) describes whether the cancer has spread to a different part of the body.
  M0 means that there is no sign that the cancer has spread. cMo(i+) means there is no sign of the cancer on physical examination, scans or x-rays. But cancer cells are present in blood, bone marrow, or lymph nodes far away from the breast cancer - the cells are found by laboratory tests M1 means the cancer has spread to another part of the body.
Clinicopathological characteristics of cancer: histopathological differentiation degree | 3 years
  Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  The histopathological differentiation is analyzed on tumor samples. The collection of a sample of the primary archival tumor and/or a sample of metastatic lesions will be requested, when available.
Clinicopathological characteristics of cancer: hormonal receptor status | 3 years
  Receptors (R) are proteins in or on cells that can attach to certain substances in the blood. Normal breast cells and some breast cancer cells have R that attach to the hormones estrogen and progesterone, and depend on these hormones to grow.
  Breast cancer cells may have one, both, or none of these R:
  * Estrogen Receptors (ER) -positive: are called ER-positive (or ER+) cancers.
  * Progesterone Receptors (PR) -positive: are called PR-positive (or PR+) cancers.
  * Hormone receptor (HR) -positive: If the cancer cell has one or both of the R above, the term hormone-receptive positive (also called hormone-positive or HR+) breast cancer may be used.
  * HR-negative: If the cancer cell has neither the ER nor the PR, it's called hormone-receptor negative (also called hormone-negative or HR-).
  The hormonal R status is analyzed on tumor samples. The collection of a sample of the primary archival tumor and/or a sample of metastatic lesions will be requested, when available.
Clinicopathological characteristics of cancer: human epidermal growth factor receptor 2 (HER2) condition | 3 years
  HER2 is a growth-promoting protein on the outside of all breast cells. Cells with higher than normal levels of HER2 are called HER2+. These cancers tend to grow and spread faster than other breast cancers, but are much more likely to respond to treatment with drugs that target the HER2 protein.
  A biopsy or surgery sample of the cancer is tested with either immunohistochemical stains (IHC) or Fluorescent in situ hybridization (FISH).
  * IHC result 0 or 1+: cancer is considered HER2-negative. These cancers do not respond to treatment with drugs that target HER2.
  * IHC result is 3+: the cancer is HER2-positive. These cancers are usually treated with drugs that target HER2.
  * IHC result is 2+: HER2 status of the tumor is not clear and is called "equivocal." HER2 status needs to be tested with FISH to clarify the result.
  HER2 is analyzed on tumor samples. The collection of a sample of the primary archival tumor and/or a sample of metastatic lesions will be requested, when available.
Clinicopathological characteristics of cancer: Ki67 proliferation index | 3 years
  Ki-67 is a protein in cells that increases as they prepare to divide into new cells. A staining process can measure the percentage of tumor cells that are positive for Ki-67. The more positive cells there are, the more quickly they are dividing and forming new cells. In breast cancer, a result of less than 10% is considered low, 10-20% borderline, and high if more than 20%.
  Ki-67 is analyzed on tumor samples. The collection of a sample of the primary archival tumor and/or a sample of metastatic lesions will be requested, when available.
Clinicopathological characteristics of cancer: BRCA1 and 2 mutations | 3 years
  BRCA1 and BRCA2 are human genes that produce tumor suppressor proteins. These proteins help repair damaged DNA and, therefore, play a role in ensuring the stability of each cell's genetic material. When either of these genes is mutated, or altered, such that its protein product is not made or does not function correctly, DNA damage may not be repaired properly. As a result, cells are more likely to develop additional genetic alterations that can lead to cancer.
  People who have inherited mutations in BRCA1 and BRCA2 tend to develop breast and ovarian cancers at younger ages than people who do not have these mutations.
  BRCA1 and 2 mutations are analyzed on whole blood samples, that are preferably collected at the enrolment visit (after signing the informed consent).
Disease-free survival (DFS) of pregnant women with breast cancer, pregnant patients after breast cancer and patients who have undergone techniques for the preservation of fertility. | 3 years
  Disease-free survival (DFS): It is defined as the time from date of initial breast cancer surgery to the date of the first documented relapse event (local, regional and/or distant) of the disease, second breast or non-breast primary tumor, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
Event-free survival (EFS) of pregnant women with breast cancer, pregnant patients after breast cancer and patients who have undergone techniques for the preservation of fertility. | 3 years
  Event-free survival (EFS): It is defined as the time from date of breast cancer diagnosis to the date of the first documented event of disease progression which excludes the potentially curative surgery, relapse (local, regional and/or distant) of the disease after the curative surgery, second breast or non-breast primary tumor, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
Progression-free survival (PFS) of pregnant women with breast cancer, pregnant patients after breast cancer and patients who have undergone techniques for the preservation of fertility. | 3 years
  Progression-free survival (PFS): It is defined as the time from the start date of a specific treatment to the documentation of disease progression on such treatment, or death due to any cause, whichever occurs first. In the event that none of the previous events were observed, censoring the last contact date will be considered.
Overall survival (OS) of pregnant women with breast cancer, pregnant patients after breast cancer and patients who have undergone techniques for the preservation of fertility. | 3 years
  Overall survival (OS): It is defined as the time from date of initial breast cancer diagnosis to the date of death due to any cause.
Correlation of the molecular profiles identified with the patients' clinicopathological and epidemiological characteristics and their disease evolution. | 3 years
Association between gestational breast cancer and a specific genotype or gene expression profile. | 3 years
Number of patients with breast cancer managed to get pregnant, spontaneously or through in vitro fertilization (IVF) methods | 3 years
  Number of patients with breast cancer managed to get pregnant, spontaneously or through in vitro fertilization (IVF) methods, considering both the patients with early disease and the patients with advanced disease.
Number of patients with breast cancer that have followed fertility preservation techniques and what type of techniques were used. | 3 years
Enumerate the potential risks of fertility preservation techniques in women with breast cancer. | 3 years
Pregnancy outcome from women diagnosed with gestational breast cancer or women with breast cancer diagnosis who became pregnant. | 3 years
Progress of the babies born from women diagnosed with gestational breast cancer or women with breast cancer diagnosis who became pregnant. | 3 years
  Regarding the live-born children, serious diseases and age until the progression is known.

OTHER OUTCOMES:
Potential relationship of clinical activity biomarkers and the probability of developing gestational breast cancer or having a relapse after the pregnancy | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Instituto Valenciano de Oncología, Valencia, España; Study Director, Study Director — Hospital Universitario Reina Sofía de Córdoba, Córdoba, España; Study Director, Study Director — Hospital Clínico Universitario de Valencia, Valencia, España; Study Director, Study Director — Centro Nacional de Epidemiología. Instituto de Salud Carlos III, Madrid, España
Locations (28):
- Spain (28):
  - Hospital Unviersitari Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Basurto, Bilbao, Bizkaia
  - Hospital Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Canary Islands
  - Complejo Hospitalario de Galicia (CHUAC), A Coruña, La Coruña
  - Hospital Universitario Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Complejo Hospitalario Reina Sofía, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud de Toledo, Toledo
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fè, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org